CLINICAL TRIAL: NCT07175896
Title: Community-based Diet Intervention for Kidney Health in Black Americans
Brief Title: Dine and DASH Into Wellness Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00118349
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Diet Interventions; Disease Prevention
Keywords: chronic kidney disease; disease prevention; pilot study; diet; DASH; dietary approaches to stop hypertension; diet intervention
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed-Start (Placebo Comparator): After randomization, the Delayed-Start group will be observed for 16 weeks with no study activity. Following the observation period, they will complete a 16-week study visit and then receive the same Kidney Health Nutrition and Cooking program that was delivered to the Immediate-Start group.
  Interventions: Behavioral: Delayed delivery of low-sodium DASH (Dietary Approaches to Stop Hypertension) diet group coaching plus hand-on cooking program
- Immediate-Start (Experimental): Each participant in the Immediate-Start arm will receive one 30-minute individual virtual session with the dietitian and advised to follow a low-sodium diet followed by 16 weekly group Kidney Health Nutrition and Cooking sessions. Didactic group sessions will occur virtually. During the ten virtual sessions, participants will be coached by a registered dietitian to follow a low-sodium DASH diet, taught to read food labels, and balance food portions. The six cooking classes will consist of hands-on instruction aimed to enhance cooking skills and help participants create nutrient-rich meals that are consistent with DASH diet principles using food staples that are common to participants' culture. Following the intervention, they will follow the DASH diet on their own for an additional 16 weeks.
  Interventions: Behavioral: Immediate delivery of low-sodium DASH (Dietary Approaches to Stop Hypertension) diet group coaching plus hand-on cooking program

INTERVENTIONS:
Behavioral: Immediate delivery of low-sodium DASH (Dietary Approaches to Stop Hypertension) diet group coaching plus hand-on cooking program — Low-sodium DASH (Dietary Approaches to Stop Hypertension) diet group coaching enhanced by cooking classes
  Arms: Immediate-Start
Behavioral: Delayed delivery of low-sodium DASH (Dietary Approaches to Stop Hypertension) diet group coaching plus hand-on cooking program — Low-sodium DASH (Dietary Approaches to Stop Hypertension) diet group coaching enhanced by cooking classes
  Arms: Delayed-Start

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of a16-week diet coaching program enhanced with cooking classes to improve adherence to the Dietary Approaches to Stop Hypertension (DASH) diet among adults who are at risk for developing chronic kidney disease.

DETAILED DESCRIPTION:
Excess cardiovascular disease (CVD) mortality among Black Americans with chronic kidney disease (CKD) is a significant US public health disparity. Compared to their White counterparts, Black adults develop kidney disease earlier in life, are 3 times more likely to develop kidney failure necessitating dialysis or kidney transplantation, and are 1.5 times more likely to die prematurely from CVD. Epidemiologic-based studies suggest that greater adherence to the Dietary Approaches to Stop Hypertension (DASH) diet improves markers of kidney function and cardiovascular outcomes in Black adults. Yet, adherence to the DASH diet is low among US adults. It is hypothesized that a 16-week culturally-tailored, dietitian-led coaching program enhanced with cooking classes will increase adherence to the DASH diet among Black adults who are at-risk for developing CKD. To inform the design of a future adequately powered clinical trial, investigators will determine the feasibility, acceptability, and preliminary efficacy of delivering a diet coaching program in community-based settings.

In this pilot trial, participants will be recruited from the local community and randomized 1:1 to receive the 16-week diet coaching program as part of an immediate-start intervention group or a delayed-start intervention group consisting of four cohorts of 12 participants. Data collection visits will occur at baseline, 16 weeks and 32 weeks. Study data will include demographic information, healthy histories, psychosocial surveys, 24-hour dietary recalls, physical measurements and laboratory data. Rates of participant recruitment, retention, group attendance and data collection will determine feasibility. Participant satisfaction ratings will determine program acceptability.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Black race
* mild to moderate chronic kidney disease, CKD (eGFR ≥ 60 ml/min/1.73m2 plus albuminuria [Stages 1 or 2] or eGFR 45-59 ml/min/1.73m2 [Stage 3a]) or normal kidney function with at least 1 of the following CKD risk factors:

  * Type 2 diabetes or pre-diabetes
  * hypertension
  * cardiovascular disease (CVD)
  * obesity
  * age 60 or older

Exclusion Criteria:

* eGFR <45 ml/min/1.73m2 (i.e., CKD stages 3b, 4, 5)
* urine dipstick consistent with nephrotic range proteinuria (>3 g)
* receiving dialysis or history of kidney transplant
* Type 1 diabetes
* pregnant, lactating or planning to become pregnant in next 6 months
* lack of internet access and videoconferencing capabilities
* planning to relocate in the next 9 months
* unable to read, write and speak in English
* participating in another research study involving diet, exercise or weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
Number of randomized participants | Up to 6 months
  Total number of participants randomized in the study during the 6 month enrollment period.

SECONDARY OUTCOMES:
Total number of study visits completed by participants | Baseline, 4 months, 8 months
Number of intervention group visits attended by participants | 4 months
Program satisfaction score | 4 months post-intervention
  Overall satisfaction score for the diet coaching program. Scored on a Likert scale of 1 (very unsatisfied) to 5 (very satisfied).
Change in DASH (Dietary Approaches to Stop Hypertension) diet score | Baseline to 16 weeks post-intervention
  A DASH diet score assesses adherence to the Dietary Approaches to Stop Hypertension diet, uses a system that gives higher points for more servings of healthy foods (fruits, vegetables, whole grains, low-fat dairy, nuts, seeds, legumes) and lower points for unhealthy foods (red meat, sweetened beverages, sodium, saturated fat). The scores are then summed, with higher overall scores indicating greater adherence to the DASH eating plan.
Change in systolic blood pressure | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference between mean clinic systolic blood pressure (mmHg) obtained at 16 weeks (end of treatment) from baseline value.
Change in diastolic blood pressure | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference between mean clinic diastolic blood pressure (mmHg) obtained at 16 weeks (end of treatment) from baseline value.
Change in random urine albumin-to-creatinine ration | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference in random urine albumin-to-creatinine ratio obtained at 16 weeks from baseline value.
Change in serum creatinine | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference in serum creatinine obtained at 16 weeks from baseline value.
Change in total cholesterol | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference in total cholesterol obtained at 16 weeks from baseline value.
Change in high-density lipoprotein | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference in high-density lipoprotein obtained at 16 weeks from baseline value.
Change in hemoglobin A1C (glycated hemoglobin) | Baseline to 16 weeks post-intervention
  Change was measured by determining the difference in hemoglobin A1C obtained at 16 weeks from baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Tyson, MD, MHS, Principal Investigator — Duke
Locations (1):
- Duke Clinical Research, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data sets that underlie results in a publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 6 months of outcome publication
Access Criteria: Qualified researchers with a sound proposal may request de-identified IPD underlying the published results. Requests should include a brief research plan/analysis plan, ethics/IRB approval or exemption, and data security procedures. Approved requesters must sign a Data Use Agreement (no re-identification, no re-distribution, analysis limited to the approved purpose, secure storage, destroy/return data at project end). Submit requests to the study PI at cs206@dm.duke.edu